CLINICAL TRIAL: NCT00822848
Title: Antiangiogenic Potentiation of Preoperative Chemoradiotherapy for High Risk Extremity Soft Tissue Sarcomas: A Phase I Study of Sorafenib With Epirubicin, Ifosfamide, Hypofractionated Radiation, and Surgery
Brief Title: Sorafenib, Epirubicin, Ifosfamide, and Radiation Therapy Followed By Surgery in Treating Patients With High-Risk Stage II or Stage III Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Christopher Ryan, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00004653; P30CA069533 (NIH); OHSU-4653; 4653; OHSU-SOL-08080-L; BAYER-OHSU-4653; CDR0000631580 (Other: NCI PDQ); NCI-2011-03738 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2009-01-14; First posted 2009-01-15 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Sarcoma
Keywords: stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma
MeSH Terms: conditions — Sarcoma | interventions — Epirubicin; Ifosfamide; Sorafenib; Immunoenzyme Techniques; Immunohistochemistry; Chemotherapy, Adjuvant; Radiotherapy, Adjuvant; Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib, Epirubicin, Ifosfamide (Experimental)
  Interventions: Drug: epirubicin hydrochloride; Drug: ifosfamide; Drug: sorafenib tosylate; Other: immunoenzyme technique; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis; Procedure: adjuvant therapy; Procedure: neoadjuvant therapy; Procedure: therapeutic conventional surgery; Radiation: hypofractionated radiation therapy

INTERVENTIONS:
Drug: epirubicin hydrochloride — I.V., days 1-3 of each cycle. Epirubicin to be omitted during cycle 2 (concomitant chemoradiation)
Drug: ifosfamide — Over 90 minutes I.V., days 1-3 of each cycle. Administered with hydration and Mesna.
Drug: sorafenib tosylate — P.O. daily beginning 2 weeks before first chemotherapy cycle, held 1 week before and after surgery.
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: adjuvant therapy — Preoperative administration has been the preference at our institution.
  Other Names: Adjuvant radiotherapy; Adjuvant chemotherapy
Procedure: neoadjuvant therapy
  Other Names: Neoadjuvant chemoradiotherapy
Procedure: therapeutic conventional surgery — Surgery should be planned for 2-4 weeks after the initiation of chemotherapy for cycle 3.
Radiation: hypofractionated radiation therapy — 28 Gy (350 centigray (cGy) x 8 fractions in 10 days) beginning at the start of cycle 2. *Boost: postoperative boost of 12 Gy (200 cGy x 6 fractions) for patients with positive surgical margins only.

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as epirubicin and ifosfamide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving chemotherapy and radiation therapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving these treatments after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This phase I trial is studying the side effects and best dose of sorafenib when given together with epirubicin, ifosfamide, and radiation therapy followed by surgery in treating patients with high-risk stage II or stage III soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine the maximum tolerated dose of sorafenib tosylate when combined with epirubicin hydrochloride, ifosfamide, and hypofractionated radiotherapy prior to surgery in patients with high-risk stage II or III soft tissue sarcoma of the extremity or body wall.

Secondary

* To examine, preliminarily, the activity of this regimen, in terms of time to local recurrence, distant disease-free survival, progression-free survival, overall survival, and histologic necrosis rate of ≥ 95%, in these patients.
* To investigate levels of tumorigenic and angiogenic markers, including phosphorylated extracellular signal-regulated kinase (p-ERK), vascular endothelial growth factor (VEGF), serum vascular endothelial growth factor receptor-2 (sVEGFR-2), and basic fibroblast growth factor (bFGF), in plasma and tumor tissue samples at baseline and during and after treatment.
* To evaluate expression of tumor proliferation and angiogenic factors, including p-ERK, vascular endothelial growth factor receptor-2 (VEGFR2) and Platelet-derived growth factor receptor (PDGFR), in tumor tissue samples as measured by Immunohistochemistry (IHC).

OUTLINE: This is a dose-escalation study of sorafenib tosylate.

Patients receive oral sorafenib tosylate* once or twice daily beginning 2 weeks before the initiation of chemotherapy and continuing until the completion of chemotherapy. Patients also receive epirubicin hydrochloride** IV and ifosfamide IV over 90 minutes on days 1-3 and pegfilgrastim subcutaneously (SC) on day 4 or filgrastim (G-CSF) (SC) daily beginning on day 4 and continuing for up to 10 days or until blood counts recover. Chemotherapy repeats approximately every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. During course 2, patients also undergo 8 fractions of external beam radiotherapy once daily between days 1-10 for a total dose of 28 Gy. Between courses 3 and 4, patients undergo surgical resection. Beginning approximately 2 weeks after surgical resection, patients with positive surgical margins undergo 6 fractions of boost external beam radiotherapy once daily for a total dose of 12 Gy.

NOTE: *Sorafenib is discontinued 1 week before surgery and resumed 1 week after surgery.

NOTE: **Epirubicin is omitted during course 2.

Plasma and tumor tissue samples are collected periodically for correlative laboratory studies. Plasma and tumor tissue samples are analyzed by ELISA for measurement of tumorigenic and angiogenic markers, including p-ERK, VEGF, sVEGFR-2, and bFGF. Tumor tissue samples are also analyzed by IHC for p-ERK, VEGFR2, phospho-VEGFR2, PDGFR, and phospho-PDGFR.

After completion of study therapy, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed soft tissue sarcoma of the upper (including shoulder) or lower (including hip) extremities or body wall
* Stage II or III disease, as defined by the following:

  * Tumor dimension > 5 cm
  * Superficial or deep tumor
  * Intermediate or high-grade disease
  * No regional lymph node involvement
  * No distant metastases
* No rhabdomyosarcoma, Ewing sarcoma, primitive neuroectodermal tumor (PNET), osteosarcoma, or gastrointestinal stromal tumor

  * Pleomorphic rhabdomyosarcoma allowed
* No known metastases

  * Patients with neurological symptoms must undergo a CT scan or MRI of the brain to exclude brain metastases

PATIENT CHARACTERISTICS:

* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Absolute Neutrophil Count (ANC) ≥ 1,500/μL
* Hemoglobin ≥ 9.0 g/dL
* Platelet count ≥ 100,000/μL
* International Normalized Ratio (INR) < 1.5 or Prothrombin Time/Partial Thromboplastin Time (PT/PTT) normal
* Creatinine ≤ 1.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 mg/dL
* Aspartate Aminotransferase/Alanine Aminotransferase (AST/ALT) ≤ 1.5 times ULN
* Left Ventricular Ejection Fraction (LVEF) ≥ 50%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception (male patients must use effective contraception for ≥ 3 months after completion of study treatment)
* No contraindications to limb-sparing surgery
* No severe peripheral vascular disease
* No concurrent uncontrolled illness including, but not limited to, the following:

  * Ongoing or active serious infection > Common Toxicity Criteria for Adverse Effects (CTCAE) grade 2
  * Symptomatic congestive heart failure
  * Unstable angina pectoris (i.e., angina symptoms at rest) or new onset angina within the past 3 months
  * Myocardial infarction within the past 6 months
  * Cardiac ventricular arrhythmia requiring anti-arrhythmic therapy
  * Psychiatric illness/social situation that would limit compliance with study requirements
* No uncontrolled hypertension (defined as systolic blood pressure > 150 mm Hg or diastolic blood pressure > 90 mm Hg, despite optimal medical management)
* No known HIV infection or chronic hepatitis B or C infection
* No thrombolic or embolic events (e.g., cerebrovascular accident, including transient ischemic attacks) within the past 6 months
* No pulmonary hemorrhage or bleeding event ≥ CTCAE grade 2 within the past 4 weeks
* No other hemorrhage or bleeding event ≥ CTCAE grade 3 within the past 4 weeks
* No serious non-healing wound, ulcer, or bone fracture
* No evidence or history of bleeding diathesis or coagulopathy
* No significant traumatic injury within the past 4 weeks
* No known or suspected allergy to sorafenib tosylate or any agent given in the study
* No condition that would impair the ability to swallow whole pills
* No malabsorption problem
* No "currently active" second malignancy other than non-melanoma skin cancer

  * Not considered to have a "currently active" malignancy if patient completed therapy AND has a < 30% risk of relapse

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy, radiotherapy, or biotherapy
* More than 4 weeks since prior major surgery
* No concurrent St. John's wort or rifampin
* No other concurrent investigational or anticancer therapy
* Concurrent anticoagulation with warfarin or heparin allowed

Ages: 15 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2009-02; Primary Completion 2012-09 (Actual); Study Completion 2013-04-30 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of sorafenib tosylate when combined with chemoradiotherapy | The first 8 weeks of therapy, but dose limiting toxicity (DLTs) will be monitored throughout the entire 22 week treatment
  The MTD is defined as the dose that produces dose limiting toxicity (DLT) in 33% of patients. Dose level escalation will be determined based on DLTs observed through the first 8 weeks of therapy, but DLTs will be monitored throughout the entire 22 week treatment course and dose de-escalation may occur if excess late DLTs are observed.
Safety | As necessary and at the discretion of the principal investigator
  As necessary and at the discretion of the principal investigator, a given dose level may be expanded by 3-6 subjects to further explore the safety of that dose level upon prior written approval of the Institutional Review Board (IRB).

SECONDARY OUTCOMES:
Time to local recurrence | From surgical resection of the primary tumor until local recurrence
  Defined as the duration of time from surgical resection of the primary tumor until local recurrence (amputated patients excluded).
Distant disease-free survival | Registration until development of distant metastatic disease or death, whichever occurs first.
  Defined as the duration of time from registration until development of distant metastatic disease or death, whichever occurs first. Subjects with stage IV disease will be censored from this analysis.
Progression-free survival | Registration to progressive disease (per RECIST)
  Defined as the duration of time from registration to progressive disease (per RECIST), local recurrence, distant metastatic disease (exclusive of stage IV subjects), or death, whichever occurs first.
Overall survival | Registration until death from any cause.
  Defined as the interval of time from registration until death from any cause.
Histologic necrosis rate of ≥ 95% | Examined for pathologic response at the time of surgery.
Levels of tumorigenic and angiogenic markers, including p-ERK, VEGF, sVEGFR-2, bFGF, in plasma and tumor tissue samples as measured by ELISA | Baseline, during, and after treatment with sorafenib plus chemoradiotherapy
Expression of tumor proliferation and angiogenic factors, including p-ERK, VEGFR2 and PDGFR, in tumor tissue samples as measured by IHC | baseline, week 2 (after sorafenib run-in), and then every 3 weeks through completion of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher W. Ryan, MD, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

REFERENCES:
- See also: NCBI PubMed Central (PMC) — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3869565/